CLINICAL TRIAL: NCT03300193
Title: The Effect of Lesion Characteristics in Magnetic Resonance Guided Focused Ultrasound Surgery (MRgFUS) on Tremor in Essential Tremor and Parkinson's Disease
Brief Title: The Effect of Lesion Characteristics in MRgFUS on Tremor in Essential Tremor and Parkinson's Disease
Acronym: MRgFUS
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Menashe Zaaroor, MD PhD, Head of Neurosurgical Department, Rambam Health Care Campus
Other Study IDs: 0162-15-RMB
Record Dates: First submitted 2016-05-29; First posted 2017-10-03 (Actual); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Tremor
Keywords: Magnetic Resonance guided Focused Ultrasound; Tremor; Essential Tremor; Parkinson's Disease
MeSH Terms: conditions — Tremor; Essential Tremor; Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tremor patients: Essential Tremor and Parkinson's Disease patients with Tremor refractory to pharmacological therapy who underwent Magnetic Resonance guided Focused Ultrasound Surgery (MRgFUS)

SUMMARY:
The study will investigate Essential Tremor and Parkinson's Disease patients who underwent Magnetic Resonance guided Focused Ultrasound Surgery (MRgFUS). We will evaluate the effect of lesion characteristics on tremor and on quality of life after the procedure as compared with the baseline prior to the procedure.

DETAILED DESCRIPTION:
The purpose of the study is to investigate the effect of lesion characteristics in ExAblate Transcranial Magnetic Resonance guided Focused Ultrasound Surgery (MRgFUS) of the Vim thalamic nucleus. Clinical measures will be used to study patients suffering from medication-refractory tremor, Essential Tremor or idiopathic Parkinson's Disease.

This study is designed as a prospective, observational, and clinical study. Assessments will be made before and after MRgFUS for; clinical tremor relief, quality of life (QoL) improvements, assessment of adverse events, and correlations of these measures with the size and shape of the lesion and the surrounding edema .

ELIGIBILITY:
Inclusion Criteria:

* Men and women, between 18 and 80 years.
* Patients who underwent the MRgFUS procedure.
* Patients who are able and willing to give consent and able to attend all study visits and Radiologic follow-up examination by MRI.
* A diagnosis of ET or Idiopathic PD as confirmed from clinical history and examination preformed by a movement disorders neurologist.
* ET patients: tremor severity score of greater than or equal to 2 in the treated hand/arm as measured by postural or action item on the Clinical Rating Scale for Tremor (CRST).
* PD patients: tremor severity score of equal or greater than 3 on either item 20 or item 21 of motor part in the Unified PD Rating Scale (UPDRS).
* Substantial disability in the performance of at least two daily activities from the disability subsection of the scales UPDRS for PD patients or CRST for ET patients.
* The patient must have a history of an unsatisfactory response to medical management. All patients will need to have tried and failed at least one drug. Alternatively, a patient may also qualify if tremor-suppressing medications are contraindicated due to a coexisting medical condition or drug allergy.
* Stable doses of all medications for 30 days prior to study entry.

Exclusion Criteria:

* Patients which have not completed the MRgFUS procedure.
* Patients which were diagnosed during the trial with additional diagnoses that can affect motor function, quality of life and symptoms of tremor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients which were diagnosed with ET or Idiopathic PD with medication refractory tremor that underwent MRgFUS procedure.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2016-05; Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Clinical Rating Scale for Tremor | 3 MONTHS
  Tremor score: In ET patients - Clinical Rating Scale for Tremor (CRST)
Motor part of Unified PD Rating Scale | 3 MONTHS
  In PD patients - Motor part of Unified PD Rating Scale (UPDRS)

SECONDARY OUTCOMES:
Quality of Life Essential Tremor Questionnaire | 3 MONTHS
  Quality of life: Quality of Life Essential Tremor Questionnaire (QUEST)
Parkinson's Disease Questionnaire | 3 MONTHS
  Parkinson's Disease Questionnaire (PDQ39)
iSeismometer application | 3 MONTHS
  For all patients: iSeismometer application for mobile phone for Assessment of tremor amplitude and frequency before and after the procedure.

OTHER OUTCOMES:
adverse events of the MRgFUS | 3 MONTHS
  Assessment of adverse events of the MRgFUS
assessment of the location of lesion on MRI | 3 MONTHS
  assessment of the location of the lesion in post procedure MRI
Size of the lesion on MRI | 3 MONTHS
  volume in mm3 of lesion in post procedure MRI
Surrounding edema on MRI | 3 MONTHS
  volume in mm3 of edema in post procedure MRI

CONTACTS AND LOCATIONS:
Overall Officials: Menashe Zaaroor, MD, DSc, Principal Investigator — Rambam Health Care Campus

IPD SHARING:
Plan to Share IPD: Yes
IPD